CLINICAL TRIAL: NCT04219137
Title: Molecular Characteristics of Gastroesophageal Adenocarcinoma (MOCHA): A Prospective Feasibility Study
Acronym: MOCHA
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 18-5663
Record Dates: First submitted 2019-12-10; First posted 2020-01-06 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Esophagogastric Adenocarcinoma
MeSH Terms: interventions — Whole Genome Sequencing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumour and blood samples will be collected for molecular characterization. Microbiome samples will also be collected for analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Localized Esophagogastric Adenocarcinoma: Patients diagnosed with gastroesophageal adenocarcinoma who will undergo surgical resection for curative intent, with or without neo-adjuvant chemotherapy or chemoradiotherapy.
  Interventions: Genetic: Molecular Profiling
- Metastatic Esophagogastric Adenocarcinoma: Patients diagnosed with de novo metastatic gastroesophageal adenocarcinoma who will undergo platinum based first line chemotherapy.
  Interventions: Genetic: Molecular Profiling

INTERVENTIONS:
Genetic: Molecular Profiling — This is a correlative study collecting biosamples to evaluate genomic characteristics and treatment outcomes of gastroesophageal adenocarcinoma.
  Other Names: Whole Genome Sequencing

SUMMARY:
Researchers are looking to further our knowledge on disease biology and treatment selection for gastroesophageal adenocarcinoma. The purpose of this study is to see how useful it is to look for changes and characteristics in your genes (molecules that contain instructions for the development and functioning of the cells) and the genes within the tumour. These characteristics may be useful in choosing treatments for patients for the future.

DETAILED DESCRIPTION:
There will be two study arms:

1. patients with suspected or diagnosed localized gastroesophageal adenocarcinoma (GEA) and
2. patients diagnosed with de novo metastatic gastroesophageal adenocarcinoma. Fresh tumour, adjacent normal tissue materials, and blood samples will be acquired and utilized to generate molecular data. Stool or rectal swab samples will also be acquired for microbiome analysis. Physiologic, quality of life, epidemiologic, frailty, and other clinical data will be systematically collected as standard of care to serve as clinical correlates for the molecular data.

Arm 1 Primary Objectives

1. Feasibility to produce a potential molecular signature in a clinically meaningful time point in patients with locally advanced GEA
2. Study the molecular characteristics of GEA in patients with localized and resectable disease and identify predictive signatures of response to induction therapy and the development of novel treatment regimens
3. To validate previously identified mutational signatures that defined subgroups of GEA

Arm 2 Primary Objectives

1. Feasibility to produce a potential molecular signature in a clinically meaningful time point for patients with advanced GEA on 1st line chemotherapy
2. Use of genotypes and genomic analyses to define therapies, and develop predictive and prognostic models
3. Assess the feasibility of prospectively identifying distinct genomic characteristics which associate with response to systemic therapy and survival

STUDY ENDPOINTS:

1. Feasibility of obtaining timely sequencing data (8-12 weeks) to guide treatment for patients progressing on 1st line treatment
2. Feasibility of using ctDNA, metabolome, immune profiling and other emerging technologies to guide treatment
3. Establish a program of personalized care for GEA patients in terms of pre-treatment assessment (Physiological and Frailty Risk Assessment, QOLQ, 4. Sarcopenia and Adiposity measurements) and treatment based on clinical-genomic correlations
4. Establishment of repository of biospecimens (tumour, blood and microbiome)
5. Establishment of robust preclinical models of GEA: PDO and PDX models
6. Assess the feasibility of using PDO models to identify drug sensitivity to guide treatment decisions

ELIGIBILITY:
Inclusion Criteria:

Arm 1:

* Patients with suspected or histologically confirmed localized gastroesophageal adenocarcinoma amenable to curative intent therapy with surgery as standard of care, either with or without induction chemotherapy or chemo radiotherapy.
* Age ≥18 years.
* Eastern Cooperative Group (ECOG) performance status 0-2

Arm 2

* Patients must have a histological or radiological diagnosis of advanced gastroesophageal cancer.
* Patient must have a tumour lesion that is amenable to a core needle biopsy as judged by a staff radiologist. A minimum of 3 x 18G good quality tumour cores must be safely obtainable under CT or US guidance. Biopsy to be completed before systemic therapy begins.
* Patients must have a measurable lesion by RECIST 1.1 in addition to the lesion that is going to be biopsied. See Section 13.1.3 for the evaluation of measurable disease. Patients with locally advanced gastroesophageal cancer with no metastatic disease who are not candidates for curative intent therapy as per part 1 of the protocol, are eligible for part 2 and are exempt from this criterion.
* Patients must be fit enough to safely undergo a tumour biopsy as judged by the investigator.
* Age ≥ 18 years.
* Eastern Cooperative Group (ECOG) performance status 0-2
* Life expectancy of greater than 90 days, as judged by the investigator.
* Patients plan to undergo systemic treatment with platinum-based chemotherapy (e.g. FOLFOX, CF, CX with or without Herceptin) as first line standard systemic palliative treatment, or as part of a first line clinical trial.
* Within 14 days of the proposed biopsy date, patients must have normal organ and marrow functions.

Exclusion Criteria:

Arm 1

* Patients who are planned for definitive chemoradiation without surgical resection will be excluded from this study.
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures.

Arm 2

* Patients with one or more contraindications to tumour biopsy according to UHN's standard biopsy procedures.
* Patients who had prior systemic treatment for advanced or metastatic gastroesophageal cancer.
* Patients who are currently on anti-cancer treatment including chemotherapy for another malignancy.
* Patients with known brain metastases are excluded from participation in this clinical study.
* Patients with advanced gastroesophageal cancer who are going to be treated with non-platinum based chemotherapy in the first line setting.
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Any condition that would, in the investigators' judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected (Arm 1) or histologically confirmed gastroesophageal adenocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-11-14 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
GEA sequencing data and molecular profiling | 2 years to recruit all patients
  Feasibility of obtaining timely sequencing data to guide treatment for patients progressing on 1st line treatment.
Establishment of GEA treatment algorithms | 2 years
  Feasibility of using ctDNA, metabolome, immune profiling and other emerging technologies to guide treatment of GEA
Establishment of personalized GEA treatment protocols | 2 years
  Feasibility to establish a program of personalized care for GEA patients in terms of pre-treatment assessment (Physiological and Frailty Risk Assessment, QOLQ, Sarcopenia and Adiposity measurements) and treatment based on clinical-genomic correlations.
GEA BioBank repository | 2 years
  Establishment of a repository of annotated, high quality blood, tumour and microbiome samples from patients with GEA. These archived specimens can be used in future research studies that aim to increase our understanding of GEA cancer and discover new ways of diagnosing and managing disease.
GEA PDO and PDX models | 2 years
  Establishment of robust patient derived tumour organoids (PDO) and Xenograft (PDX) models, and then assess feasibility of using models to identify drug sensitivity to guide treatment decisions.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Elimova, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada